CLINICAL TRIAL: NCT00265525
Title: Evaluation of a Web-Based Intervention to Promote Physical Activity in Patients With Heart Disease: A Randomize Control Trial
Brief Title: Evaluation of a Web-based Intervention to Promote Physical Activity in Patients With Heart Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Robert Reid/Principal Investigator, University of Ottawa Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HBR 4855
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Randomized Control Trial; Exercise Intervention; Prevention; Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardio fit (Experimental)
  Interventions: Behavioral: CardioFit
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: CardioFit — CardioFit is a 26-week tailored web-based physical activity coaching service for individuals with Coronary Artery Disease (CAD). It has been designed to help patients develop personalized exercise programs based on their medical history, personal goals and preferences. Access to Cardio-fit is through a secured website. The cardio-fit website contains physical activity advice and heart health educational information. Each patient is assigned an on-line coach, whose role is to assist in creating safe an effective physical activity program, and to answer any questions that patients may have throughout the program.
  Arms: Cardio fit

SUMMARY:
A randomized control trial (RCT) is planned to evaluate a web-based intervention (CardioFit) against usual care in increasing physical activity levels in patients with Coronary Artery Disease (CAD). We hypothesize that compared to usual care, participants in CardioFit will; a) have increased physical activity levels, b) will have a higher health-related quality of life at measurement dates and, c) will have greater improvements in psychosocial predictors.

DETAILED DESCRIPTION:
Most existing cardiac rehabilitation programs have little ability to expand participation using traditional delivery models that emphasize supervised, facility-based programs. Futhermore, facility based programs to promote physical activity behavior in patients with coronary artery disease (CAD) are limited in their impact because most patients are unwilling to travel more than 30-40 minutes to participate in a program. CardioFit is an off-site, 26 week web-based physical activity coaching service for people with heart disease. Within the CardioFit program, patients will be assigned to an on-line "coach" and receive customized exercise programs based on their medical history, personal goals and preferences. A randomized control trial (RCT) is planned to evaluate the effectiveness of the web-based intervention at increasing physical activity levels against usual care in patients with CAD.

This study is in the third phase of a three-phase research program to examine interventions to promote physical activity for the secondary prevention of Cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80 years
* English Proficiency
* Internet Access (home or work)
* Documented CAD (most recent cardiac diagnosis); documented Myocardial Infarction (MI), successful PCI procedure

Exclusion Criteria:

* Patient intends to enroll in structured cardiac rehabilitation
* Hospitalization for Coronary Artery Bypass (CABG)
* Hospitalization for diagnostic procedure not associated with previously documented MI
* Patient coming back to hospital for planned staged PCI within 6 months
* Cardiac transplantation
* Presence of, or hospitalization for defibrillator implant
* Hospitalization for pacemaker implantation
* Unresolved unstable angina &/or hospitalization for angina (without MI or PCI)
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
* Neuromuscular, musculoskeletal or rheumatoid disorders that are exacerbated by exercise
* Other uncontrolled metabolic conditions (e.g. diabetes)
* Chronic infectious diseases such as mononucleosis, hepatitis, AIDS
* Acute systematic illness or fever
* Uncontrolled tachycardia (<120 bpm)
* Uncompensated congestive heart failure (&/or NYHA Class III, or IV)
* 3rd degree AV block without pacemaker
* Active pericarditis or myocarditis
* Recent embolism
* Suspected or known AAA aneurysm > 4cm
* Uncontrolled hypertension (SBP > 200; DBP > 110)
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Physical activity: measured at baseline (day of hospital discharge), 6 months and 12 months via: | Baseline, 6 and 12 months

SECONDARY OUTCOMES:
Measured at baseline, 6 months, and 12 months via follow-up questionnaire: | Baseline, 6 and 12 months
Recurrent cardiac events | Baseline, 6 and 12 months
Barriers | Baseline, 6 and 12 months
Task Self-efficacy | Baseline, 6 and 12 months
Outcome expectations | Baseline, 6 and 12 months
Social Support | Baseline, 6 and 12 months
Perceived environment | Baseline, 6 and 12 months
Heart disease specific quality of life | Baseline, 6 and 12 months
Use of secondary prevention medications | 6 and 12 months
Pedometer (9days) | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Reid, PhD, Principal Investigator — University of Ottawa Heart Institute, Prevention and Rehabilitation Centre; Andrew Pipe, C.M, MD, Study Chair — University of Ottawa Heart Institute, Prevention and Rehabilitation Centre; Louise Morrin, MBA, B.Sc., Study Chair — University of Ottawa Heart Institute, Prevention and Rehabilitation Centre
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Unversity of Ottawa Heart Institute, Ottawa, Ontario

REFERENCES:
- [Derived] Reid RD, Morrin LI, Beaton LJ, Papadakis S, Kocourek J, McDonnell L, Slovinec D'Angelo ME, Tulloch H, Suskin N, Unsworth K, Blanchard C, Pipe AL. Randomized trial of an internet-based computer-tailored expert system for physical activity in patients with heart disease. Eur J Prev Cardiol. 2012 Dec;19(6):1357-64. doi: 10.1177/1741826711422988. Epub 2011 Sep 8. PMID 21903744
- [Derived] Reid RD, Morrin LI, Higginson LA, Wielgosz A, Blanchard C, Beaton LJ, Nelson C, McDonnell L, Oldridge N, Wells GA, Pipe AL. Motivational counselling for physical activity in patients with coronary artery disease not participating in cardiac rehabilitation. Eur J Prev Cardiol. 2012 Apr;19(2):161-6. doi: 10.1177/1741826711400519. Epub 2011 Feb 21. PMID 21450579
- See also: University of Ottawa Heart Institute website — http://www.ottawaheart.ca/